CLINICAL TRIAL: NCT03255057
Title: A Prospective, Multi-Center, Randomized, Controlled, Pivotal Trial to Validate the Safety and Efficacy of the Hemolung® Respiratory Assist System for COPD Patients Experiencing an Acute Exacerbation Requiring Ventilatory Support
Brief Title: Extracorporeal CO2 Removal With the Hemolung RAS for Mechanical Ventilation Avoidance During Acute Exacerbation of COPD
Acronym: VENT-AVOID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment post COVID-19 pandemic
Sponsor: Alung Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HL-CA-5000
Record Dates: First submitted 2017-08-09; First posted 2017-08-21 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Acute Exacerbation of COPD

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, randomized, controlled, two-arm, open-label, adaptive, two-strata, pivotal trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the interventional device and treatment, the study participants, care providers, and investigators will not be masked. However, an independent Clinical Endpoint Committee will be masked for adjudication of the primary endpoint and serious adverse events. An independent Data and Safety Monitoring Board will make study continuation recommendations based on the statistical analysis plan and the overall safety and efficacy endpoints without masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Hemolung plus SOC IMV (Experimental): Low-flow ECCO2R with the Hemolung Respiratory Assist System as an alternative or adjunct to standard-of-care (SOC) invasive mechanical ventilation (IMV)
  Interventions: Device: Hemolung Respiratory Assist System; Device: Invasive mechanical ventilation
- SOC IMV (Active Comparator): Standard-of-care (SOC) invasive mechanical ventilation (IMV) alone
  Interventions: Device: Invasive mechanical ventilation

INTERVENTIONS:
Device: Hemolung Respiratory Assist System — Treatment with a medical device called the Hemolung RAS. The Hemolung RAS includes three components: the Hemolung Controller, the Hemolung Cartridge, and the Hemolung Catheter. The intervention is use of the Hemolung RAS to provide partial lung support for acute hypercapnic lung failure by filtering carbon dioxide from venous blood using a central venous catheter through which venous blood is pumped at flows of 350-550 milliliters per minute to and from an external circuit containing a hollow fiber membrane blood gas exchanger (with heparin-coated fibers) integrated with a centrifugal pump.
  Other Names: Low-flow extracorporeal carbon dioxide removal; ECCO2R; Hemolung RAS; Hemolung; Respiratory dialysis; Lung dialysis
  Arms: Hemolung plus SOC IMV
Device: Invasive mechanical ventilation — Lung support for acute lung failure applied with a mechanical ventilation device that uses positive pressure to mechanically inflate the lungs and facilitate exhalation via an endotracheal tube or tracheotomy.

SUMMARY:
This study evaluates the safety and efficacy of using the Hemolung RAS to provide low-flow extracorporeal carbon dioxide removal (ECCO2R) as an alternative or adjunct to invasive mechanical ventilation for patients who require respiratory support due to an acute exacerbation of Chronic Obstructive Pulmonary Disease (COPD). It is hypothesized that the Hemolung RAS can be safely used to avoid or reduce time on invasive mechanical ventilation compared to COPD patients treated with standard-of-care mechanical ventilation alone. Eligible patients will be randomized to receive lung support with either the Hemolung RAS plus standard-of-care mechanical ventilation, or standard-of-care mechanical ventilation alone.

DETAILED DESCRIPTION:
The Hemolung RAS provides low-flow ECCO2R using a single, 15.5 French dual-lumen catheter inserted percutaneously in the femoral or jugular vein. Low-flow ECCO2R offers an alternative or supplement to invasive mechanical ventilation (MV) for patients suffering from acute, reversible, hypercapnic respiratory failure. In contrast to invasive MV, low-flow ECCO2R provides partial ventilatory support independently of the lungs. The rationale for this study is that low-flow ECCO2R with the Hemolung RAS can be used to provide supplemental CO2 removal in COPD patients experiencing acute hypercapnic respiratory failure to either avoid or reduce time on invasive MV. In this patient population, avoidance or reduced time on invasive MV may have significant clinical benefit in reducing the many complications associated with invasive MV. The major complication risks of low-flow ECCO2R are associated with central venous catheterization and the need for anticoagulation during treatment. This study is designed to evaluate the safety and efficacy of Hemolung RAS plus standard-of-care as compared to standard-of-care alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 40 years
2. Confirmed diagnosis of underlying COPD or ACOS (Asthma-COPD Overlap Syndrome)
3. Experiencing acute hypercapnic respiratory failure
4. Informed consent from patient or legally authorized representative
5. Meets one of the three following criteria:

   1. Is at high risk of requiring intubation and invasive mechanical ventilation (MV) after at least one hour on NIV due to one or more of the following:

      * Respiratory acidosis (arterial pH <= 7.25) despite NIV
      * Worsening hypercapnia or respiratory acidosis relative to baseline blood gases
      * No improvement in PaCO2 relative to baseline blood gases and presence of moderate or severe dyspnea
      * Presence of tachypnea > 30 breaths per minute
      * Intolerance of NIV with failure to improve or worsening acidosis, dyspnea or work of breathing

      *OR*
   2. After starting NIV with a baseline arterial pH ≤ 7.25, shows signs of progressive clinical decompensation manifested by decreased mental capacity, inability to tolerate NIV, or increased or decreased respiratory rate in setting of worsened or unchanged acidosis.

      *OR*
   3. Currently intubated and receiving Invasive MV, meeting both of the following:

      * Intubated for ≤ 5 days (from intubation to time of consent), AND
      * Has failed a spontaneous breathing trial OR is deemed not suitable for a spontaneous breathing trial (SBT) OR is deemed not suitable for extubation

Exclusion Criteria:

1. DNR/DNI order
2. Hemodynamic instability (mean arterial pressure < 60 mmHg) despite infusion of vasoactive drugs
3. Acute coronary syndrome
4. Current presence of severe pulmonary edema due to Congestive Heart Failure
5. PaO2/FiO2 < 120 mmHg on PEEP >/= 5 cmH2O
6. Presence of bleeding diathesis or other contraindication to anticoagulation therapy
7. Platelet count >= 100,000/mm3 not requiring daily transfusions to maintain platelet count above 100,000/mm3 at time of screening
8. Hemoglobin >= 7.0 gm% not requiring daily transfusions to maintain hemoglobin count above 7.0 gm% at time of screening, and no active major bleeding
9. Unable to protect airway (e.g. unable to generate cough or clear secretions) or significant weakness or paralysis of respiratory muscles due to causes unrelated to acute exacerbation of COPD
10. Cerebrovascular accident, intracranial bleed, head injury or other neurological disorder likely to adversely affect ventilation or airway protection.
11. Hypersensitivity to heparin or history of previous heparin-induced thrombocytopenia (HIT Type II)
12. Presence of a significant pneumothorax or bronchopleural fistula
13. Current uncontrolled, major psychiatric disorder
14. Current participation in any other interventional clinical study
15. Pregnant women (women of child bearing potential require a pregnancy test)
16. Neutropenic (absolute neutrophil count < 1,00mm3, not transient) related to the presence or treatment of a malignancy; recent bone marrow transplant (within prior 8 months); current, uncontrolled AIDS.
17. Fulminant liver failure
18. Known vascular abnormality or condition which could complicate or prevent successful Hemolung Catheter insertion
19. Terminal patients not expected to survive current hospitalization
20. Requiring continuous home ventilation via a tracheostomyy
21. Any disease or condition that, in the judgment of the investigator, either places the subject at undue risk of complications from the Hemolung RAS device, or may reduce the subject's likelihood of benefitting from therapy with the Hemolung RASr

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-02-18 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
The amount of time in the first five days following randomization that a patient is free of Invasive MV and alive | 5 days
  Statistically analyzed as Ventilator-Free Days during the 5 days from randomization (VFD-5)

SECONDARY OUTCOMES:
Physiologic benefit | Time to extubation from first intubation up to 60 days from randomization
  Based on blood gases and concomitant ventilation parameters
Avoidance of intubation | Within 60 days from randomization
  Incidence of subjects who did not require intubation at any time during their primary hospital admission for the exacerbation for which they were enrolled in the study.
Ability to communicate by speaking | Randomization to end of treatment or 14 days, whichever is sooner
  Number of days from randomization to end of treatment (end of Invasive MV in Control Arm and end of Hemolung treatment in Investigational Arm) subject is able to communicate by speaking
Ability to eat and drink orally | Randomization to end of treatment or 14 days, whichever is sooner
  Number of days from randomization to end of treatment (end of Invasive MV in Control Arm and end of Hemolung treatment in Investigational Arm) subject is able to eat and drink orally
ICU Mobility | Randomization to end of treatment or 14 days, whichever is sooner
  Ability of subject to mobilize in bed and out of bed while in Intensive Care as assessed using ICU Mobility Score (IMS)
Daily dose of sedatives, analgesics, and paralytics while in ICU | From randomization to ICU discharge up to 60 days from randomization
  A qualify of life measure for subjects while in ICU measured by reported concomitant medications while in ICU.
Incidence of new tracheotomies | Within 60 days from randomization
  Incidence of new tracheotomies
Adverse events | Within 60 days from randomization
  All Serious Adverse Events (SAE) from randomization to 60 days and non-serious adverse events from randomization to ICU discharge or 30 days, whichever is sooner (adjudicated by the Clincal Events Committee)
All-cause in-hospital mortality | Within 60 days from randomization
  Subject death from any cause while still admitted to hospital for the acute exacerbation for which they were enrolled in the study.
All-cause (health-related) mortality at 60 days from randomization | Within 60 days from randomization
  Incidence of health-related deaths at 60 days from randomization, regardless of subject location at time of death.
Incidence of failed extubations | Within 60 days from randomization
  Incidence of re-intubation within 48 hours of extubation for original exacerbation

OTHER OUTCOMES:
Time to ICU discharge | From ICU admission to discharge up to 60 days from randomization
  Time from ICU admission to ICU discharge for initial exacerbation for which the subject was enrolled for subjects surviving to discharge
Time to hospital discharge | From hospital admission to discharge up to 60 days from randomization
  Time from hospital admission to hospital discharge for initial exacerbation for which the subject was enrolled for subjects surviving to discharge
Time on ventilatory support | Randomization to end of Hemolung an Invasive MV for initial exacerbation up to 60 days from randomization
  Total time on Hemolung and/or Invasive MV support for initial exacerbation
VFD-30 | Randomization to Day 30
  Ventilator-free days from randomization to 30 days from randomization
SOFA Score | From randomization to 24 hours after end of investigational treatment (Investigational Arm) or first extubation (Control Arm) up to a maximum of 14 days
  Sequential Organ Failure Assessment Score from randomization to 24 hours after end of treatment
Dyspnea | From randomization to 24 hours after end of investigational treatment (Investigational Arm) or first extubation (Control Arm) up to a maximum of 14 days
  A quality of life measure for subjects while in ICU measured with a Visual Analog Score
ICU Delirium | From randomization to 24 hours after end of investigational treatment (Investigational Arm) or first extubation (Control Arm) up to a maximum of 14 days
  A quality of life measure for subjects while in ICU measured with the Confusion Assessment Measure for ICU (CAM-ICU) score
Incidence of DNI/DNR/Comfort care requests post-randomization | From randomization to 60 days from randomizaiton
  Incidence of DNI/DNR/Comfort care requests post-randomization
Incidence of hospital readmissions | From randomization to 60 days from randomizaiton
  Number of new hospital admissions after hospital discharge for original exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hill, MD, Principal Investigator — Tufts University Medical Center
Locations (32):
- United States (32):
  - UC Davis Medical Group, Sacramento, California
  - Denver Health Medical Center, Denver, Colorado
  - Christiana Care Health System, Newark, Delaware
  - University of Florida - Health Shands, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - WellStar Kennestone Regional Medical Center, Marietta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Lexington VA Healthcare, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - LSU Health Shreveport, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Minneapolis Heart, Minneapolis, Minnesota
  - Rutgers-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Northwell Health, New Hyde Park, New York
  - New York Presbyterian Hospital/Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - UT Erlanger, Chattanooga, Tennessee
  - Memphis VA Medical Center, Memphis, Tennessee
  - UT McGovern Medical School Memorial Hermann, Houston, Texas
  - Baylor Scott and White Memorial Hospital, Temple, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Health Care Services, Falls Church, Virginia

REFERENCES:
- [Background] Burki NK, Mani RK, Herth FJF, Schmidt W, Teschler H, Bonin F, Becker H, Randerath WJ, Stieglitz S, Hagmeyer L, Priegnitz C, Pfeifer M, Blaas SH, Putensen C, Theuerkauf N, Quintel M, Moerer O. A novel extracorporeal CO(2) removal system: results of a pilot study of hypercapnic respiratory failure in patients with COPD. Chest. 2013 Mar;143(3):678-686. doi: 10.1378/chest.12-0228. PMID 23460154
- [Derived] Duggal A, Conrad SA, Barrett NA, Saad M, Cheema T, Pannu S, Romero RS, Brochard L, Nava S, Ranieri VM, May A, Brodie D, Hill NS; VENT-AVOID Investigators. Extracorporeal Carbon Dioxide Removal to Avoid Invasive Ventilation During Exacerbations of Chronic Obstructive Pulmonary Disease: VENT-AVOID Trial - A Randomized Clinical Trial. Am J Respir Crit Care Med. 2024 Mar 1;209(5):529-542. doi: 10.1164/rccm.202311-2060OC. PMID 38261630
- [Derived] Stokes JW, Gannon WD, Rice TW. Extracorporeal Carbon Dioxide Removal or Extracorporeal Membrane Oxygenation: Why Should We Care? Crit Care Med. 2021 May 1;49(5):e546-e547. doi: 10.1097/CCM.0000000000004844. No abstract available. PMID 33854019